CLINICAL TRIAL: NCT05594056
Title: Transorbital Ultrasound Measurement of Optic Nerve Sheath Diameter Between Pregnant Women With Severe Preeclampsia and Normal Gestations. Prospective, Controlled Trial.
Brief Title: Transorbital Ultrasound of Optic Nerve Sheath Diameter Between Healthy Pregnant Women and Those With Severe Preeclampsia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Chairman of Research Department, Saint Thomas Hospital, Panama
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-600
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Preeclampsia Severe
Keywords: Severe preeclampsia; Optic nerve sheet; Intracranial pressure
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: A transorbital ultrasound to measure the optic nerve sheet will be performed in patients with severe preeclampsia and then compared with normal controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preeclampsia (Experimental): Patients with severe preeclampsia and gestational age between 34-40 weeks.
  Interventions: Procedure: Transorbital ultrasound of the optic nerve sheet
- Control (Active Comparator): Patients with normal gestations between 34-40 weeks.
  Interventions: Procedure: Transorbital ultrasound of the optic nerve sheet

INTERVENTIONS:
Procedure: Transorbital ultrasound of the optic nerve sheet — Measurement of the optic nerve sheet with a linear transducer (7,5 MHz).

SUMMARY:
The neurological alterations associated with preeclampsia depend on cerebral autoregulation, a theory that outlines the mechanisms by which the nervous system controls cerebral perfusion. However, with the loss of autoregulation, increased blood flow, edema and eventually increased intracranial pressure are triggered and may be translated into neurological manifestations such as symptoms of vasospasm, one of the criteria for severity in preeclampsia.

Nervous system manifestations frequently found in preeclampsia are headache, blurred vision, scotomas and hyperreflexia. Although uncommon, temporary blindness (lasting a few hours to a week) may also accompany severe preeclampsia and eclampsia.

The optic nerve, as part of the central nervous system, is surrounded by cerebrospinal fluid and dura mater, which forms the optic nerve sheath. Due to the connection with the intracranial subarachnoid space, the diameter of the optic nerve sheath is influenced by variations in cerebrospinal fluid pressure. Increased intracranial pressure is transmitted to the subarachnoid space surrounding the optic nerve, causing its expansion.

Recent studies suggest that an optic nerve sheath diameter greater than 5 mm correlates 100% with ICP (intracerebral pressure) greater than 20 mm Hg. Due to the simple nature of the test and the limited time required to perform it, it is an ideal non-invasive test to assess changes in mental status, severe headache, and to take the necessary measures aimed at reducing intracranial pressure.

The diagnosis of elevated intracranial pressure is challenging and critical, because early recognition and treatment are essential to prevent brain damage or death since preeclampsia with severe data remains one of the most frequent complications in our institution.

These values are not taken from the obstetric population, so this study proposes the description of a standard value for the pregnant population. There are few studies that describe a value to help us define cases of this pathology and correlate it with the signs and symptoms of severity in patients with preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15-44 years.
* Gestational age between 34-40 weeks of gestation.

Exclusion Criteria:

* Eye disease (Glaucoma, diabetic neuropathy, optic neuritis).
* Nervous disorders.
* Psychiatric disorders
* Diabetes

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheet measurement | 24 hours
  The diameter of the optic nerve sheath was measured three millimeters behind the eyeball, and one axis perpendicular to the optic nerve. Three measurements were taken in each eye. The resulting six measurements were averaged to give a mean of the optic nerve sheet measurement, to minimize measurement variability.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Study Chair — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas H, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No